CLINICAL TRIAL: NCT06116942
Title: Repetitive Transcranial Magnetic Stimulation for Enhancing Brain Computer Interphase-induced Plasticity in Stroke: a Crossover Design
Brief Title: Magnetic Brain Stimulation and Computer-based Motor Training for Rehabilitation After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Collaborators: University of Halle Medical Faculty (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Neurotech Stroke; DE-23-00014797 (Registry Identifier: Bundesinstitut für Arzneimittel und Medizinprodukte)
Record Dates: First submitted 2023-09-27; First posted 2023-11-03 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Chronic Stroke
Keywords: Transcranial Magnetic Stimulation; Intermittent Theta Burst Stimulation; Brain-Computer Interface; Rehabilitation; EEG; MRI; Molecular changes; Brain plasticity; Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled cross-over factorial single-blind mono-center trial with 2 arms (active stimulation-placebo stimulation | placebo stimulation-active stimulation).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation - Placebo stimulation (Experimental): Participants will undergo a 2 intervention periods. The first intervention period will consist of a 2-week course of rTMS followed by BCI-mediated training. This intervention will be succeeded by a 4-week washout period to mitigate any carry-over effects. The second intervention period will entail 2 weeks of sham rTMS followed by BCI-mediated training.
  Interventions: Device: Active rTMS; Device: Sham rTMS
- Placebo stimulation - Active stimulation (Experimental): Participants will undergo the same interventions as the first arm but delivered in inverse order. The first intervention period will consist of 2 weeks of sham rTMS followed by BCI-mediated training. The second intervention period will entail 2 weeks of rTMS prior to BCI-mediated training and will start after a 4-weeks washout period.
  Interventions: Device: Active rTMS; Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — The Transcranial Magnetic Stimulation will consist of placing a figure-of-eight shape coil of wire over the head of the participants. Then, a brief electric current will pass through the coil, inducing a magnetic field capable of stimulating neurons located beneath the coil. For the active coil, the maximal stimulation intensity is reached beneath the center of the coil.
  In the present study, the intermittent theta-burst protocol will be implemented. This protocol is expected to modulate the excitability of the brain, priming it for a stronger activation of the motor-related brain areas engaged during brain-computer interface-based training. The structural MRI of each participant will be used to guide neuronavigation towards ipsilesional motor areas.
  Other Names: Intermittent Theta Burst Stimulation; Repetitive Transcranial Magnetic Stimulation; iTBS
Device: Sham rTMS — To implement a placebo stimulation, a sham coil will be used to deliver the same stimulation protocol. The sham coil is identical in dimensions and weight to the active coil but produces a diminished magnetic field. For the sham coil, the stimulation intensity is minimal beneath the center of the coil, the same area with the highest intensity during stimulation with an active coil. The structural MRI scan of each participant will be used to guide neuronavigation towards the same area where the active stimulation was applied.
  Other Names: Placebo Intermittent Theta Burst Stimulation; Placebo Repetitive Transcranial Magnetic Stimulation; Sham iTBS

SUMMARY:
The goal of the present clinical trial is to explore whether an innovative technology-based approach can help individuals who have had a stroke and can no longer move their hands with ease. Our approach consists of a combination of two technologies: Transcranial Magnetic Stimulation (TMS) and a Brain-Computer Interface (BCI). The former entails the application of magnetic fields over the head to stimulate the brain preparing it for a better ability to produce movement. The latter consists of measuring brain activity to personalize a type of computer-based training that is designed to increase communication between the brain and the muscles.

DETAILED DESCRIPTION:
Aims of the study:

1. to provide preliminary evidence of the effect of rTMS (repetitive Transcranial Magnetic Stimulation) on brain-computer interface (BCI)-mediated plasticity on individuals with hemiparesis after stroke
2. Measure adherence and withdrawal rates of the present protocol for informing a future large-scale randomized controlled trial

The active stimulation (rTMS) consists of an intermittent theta burst (iTBS) protocol whereas the placebo condition encompasses rTMS stimulation delivered with a Sham coil (Sham).

Procedures:

The study will entail 25 sessions. The study is composed of six different types of sessions in a crossover design:

1. Screening session (day 1): Includes the informed consent form signature, enrollment and BCI calibration
2. Before-treatment and after-treatment sessions (day 2, 13, 14 and 25) include the recording of EEG and MRI data, as well as the application of tests and questionnaires for evaluation of motor function
3. Daily visit with blood draw sessions (days 3, 12, 15 and 24): consist of the delivery of active or sham rTMS followed by BCI training preceded and followed by a blood draw.
4. Daily visit sessions without a blood draw (days 4 to 11 and 16 to 23): consist of the delivery of active or sham rTMS followed by BCI training.

After a screening session (day 1), the clinical study begins. The period I of the study begins with a before-treatment session (day 2). Then, the intervention (rTMS or sham followed by BCI training) is delivered during 10 daily visits over a 2-week period excluding weekends (days 3 to 12). Within the daily visits, there are 2 daily visits with blood draws (days 3 and 12) and the rest do not include any blood draws (days 4 to 11). Then, an after-treatment session takes place (day 13).

After period I, a washout period of 4 weeks takes place. No measurements or training are required during this time. In Period II of the study, the session flow is repeated except for the screening session. Therefore, period II includes a before-treatment session (day 14), 10 daily visits (days 15 to 24), with 2 daily visits that include blood draws (days 15 and 24), and an after-treatment session (day 25).

Research questions:

1. Does rTMS promote better motor recovery after BCI training in comparison to sham?
2. Can rTMS propitiate stronger effects on neural physiology after BCI training in comparison with sham?
3. Is there an association between behavioral and physiological changes after the proposed intervention?
4. What is the adherence and withdrawal rate and reason for withdrawal of the proposed study design and procedures?
5. Is there an association between brain structures associated with motor function at baseline and the changes observed after rTMS?
6. Can applying rTMS have a better effect on self-perceived motor performance in daily activities in comparison to Sham?
7. Are serum molecular markers of plasticity and neural turnover modulated by rTMS?

Hypotheses:

1. A higher increase in motor performance will be observed after the rTMS-BCI in comparison with sham-BCI. The motor performance will be assessed as Fugl-Meyer Assessment for upper extremity score as the primary outcome measure; and as the Jebsen Taylor hand function test and BCI accuracy as the secondary outcome measures
2. Higher physiological changes will be observed after rTMS-BCI in comparison with sham-BCI. The electrophysiological changes will be assessed as Motor evoked potentials, as primary outcome measured; and as motor-related cortical potentials, Event-Related Desynchronization and functionalMagnetic Resonance Imaging changes as secondary outcome measures
3. Behavioral and physiological changes will be associated
4. Changes in structural MRI will be associated with behavioral outcome measures after rTMS-BCI and sham-BCI. Structural MRI will be assessed as Fractional Anisotropy changes, as a primary outcome measure; and voxel-based morphometry as a secondary outcome measure
5. Individuals will have a higher perceived improvement in activities of daily living, measured as higher scores in the Upper extremity motor activity log (UE-MAL) and the first and last items of the Stroke impact scale (SIS) questionnaire after rTMS-BCI in comparison with sham-BCI
6. The increase in Brain-Derived Neurotrophic Factor (BDNF) will be higher after rTMS-BCI in comparison with after sham-BCI and an association between BDNF levels and behavioral markers of motor recovery will exist

As an exploratory analysis, the investigators will inspect preliminary evidence of the effects of the stimulation by verifying changes in serological markers of neuronal plasticity and turnover.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a subcortical stroke at least 6 months before the initiation of the trial and confirmed with magnetic resonance imaging (MRI) or computed tomography
2. Present moderate to severe hemiparesis in an upper limb
3. Language comprehension as well as visual and auditory perception sufficient to engage in Brain Computer Interface training
4. Age from 20 to 80 years old
5. Clear consciousness and stable vital signs
6. Eligible for MRI, EEG, BCI and TMS methods

Exclusion Criteria:

1. Drug abuse or recent changes in medications that may alter the central nervous system when the measurements begin or during the measurements (e.g., benzodiazepines, serotoninergic and dopaminergic agents)
2. History of seizure
3. Bone, joint and muscle diseases
4. Peripheral neuropathy or other neurological or psychiatric diseases (including, tinnitus, migraine, or mood disorders with the exception of minimal, mild, and moderate depression, reflected as a Beck depression scale score lower than 29).
5. Strong cognitive deficits (including speech, attention, hearing, vision, sensation or intelligence deficits) reflected as a Montreal Cognitive Assessment (MoCA) score lower or equal to 24
6. Lesions in the upper extremities
7. Bone, joint and muscle diseases
8. Severe spasticity (higher than 3) or pain in the upper limb and affecting wrist extension
9. Contraindications of undergoing TMS examinations: history of seizures, history of epilepsy, unclear unconsciousness, migraines or metals on the head
10. Contraindications for MRI: metals in the body, metallic prosthetics or claustrophobia
11. Participation in other interventional trials using BCI or rTMS within less than 6 months ago
12. Participation in another interventional clinical trial
13. Suspected lack of compliance
14. Pregnant or nursing women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-08 (Estimated); Primary Completion 2026-09-19 (Estimated); Study Completion 2027-09-19 (Estimated)

PRIMARY OUTCOMES:
Motor-evoked potential (MEP) parameters | Measured two times per day, at the days: 3-12 and 15-24. The first measurement is performed immediately before the rTMS-BCI intervention and the second immediately after the rTMS-BCI intervention.
  An MEP is the electromyography response to a single TMS pulse delivered over the motor cortex, over the representation of multiple muscles. MEP changes will be evaluated with a mixed effects model. mixed-effects model. The model will consider the Patient, Period, Treatment (stimulation type) and Session number. The Period*Treatment interaction will be verified to detect carry-over effects. The investigators expect to observe a main effect of Treatment and Session number.
Fugl-Meyer upper extremity assessment of sensorimotor function | Measured one time at day, at the days: 2, 13, 14, and 25.
  Quantitative evaluation of motor, balance, sensation and joint functions. The sums of values recorded before and after the stimulation periods will be fed into an unpaired sample t-test to evaluate carryover effects whereas the differences observed between recordings before and after the stimulation will be fed into an unpaired sample t-test for the evaluation of initial evidence of the effect of rTMS.
Event-related desynchronization (ERD) | Measured one time per day, at the days: 2, 13, 14, and 25.
  Electroencephalography (EEG) will be recorded during a cued motor task. This data will be used to calculate event-related de-synchronization, defined as the difference in signal power in the miu (8-12 Hz) and beta bands (13-30 Hz) between a baseline period prior to the cue and a post-cue period. Changes in ERD will be evaluated with permutation-based statistics.

SECONDARY OUTCOMES:
Brain-Computer Interface accuracy | Measured one time per day, at days 3-12 and days 15-24.
  Ratio of correct trials over the total number of trials, as a proxy of performance during brain-computer interface based training. BCI accuracy will be evaluated with a mixed-effects model. mixed-effects model. The model will consider the Patient, Period, Treatment (stimulation type) and Session number. The Period*Treatment interaction will be verified to detect carry-over effects. The investigators expect to observe a main effect of Treatment and Session number.
Task-related functional Magnetic Resonance Imaging (t-fMRI) | Measured one time per day, at the days 2, 13, 14, and 25.
  fMRI will be acquired during a motor task. The fMRI acquired during the task will be used to evaluate blood-oxygen-level-dependent (BOLD) signal changes after the active stimulation over the motor areas: premotor cortex (PMC), motor cortex (M1), supplementary motor area (SMA), cerebellum and basal ganglia; and this change will be compared with the change after placebo stimulation. In addition, the investigators will explore whether changes in BOLD signal in areas involved in BCI training can be observed after active stimulation, reflecting a potential enhancement of BCI effects. Changes in fMRI will be evaluated with a mixed-effects model in a whole-brain analysis.
Jebsen-Taylor Hand Function Test | Measured one time per day, at the days 2, 13, 14, and 25.
  Clinical assessment of hand function that consists of 7 tasks: staking checkers, feeding, manipulating and lifting objects, writing, and page-turning. The sums of values recorded before and after the stimulation periods will be fed into an unpaired sample t-test to evaluate carryover effects whereas the differences observed between recordings before and after the stimulation will be fed into an unpaired sample t-test for the evaluation of initial evidence of the effect of rTMS.
Diffusion-based tractography | Measured one time per day, at the days 2, 13, 14, and 25.
  Evaluation of fractional anisotropy (FA) as a proxy of white matter changes. Diffusion-weighted images will be used to used to calculate FA. FA reflects the deviation of random diffusion of water molecules in a voxel. Analysis of effects in diffusion will be carried out at the whole brain level and using contrast weights in a flexible factorial design with multiple groups of subjects.
Movement-related cortical potential amplitude | Measured one time per day, at the days 2, 13, 14, and 25.
  Electroencephalography (EEG) will be recorded during a cued-motor task. The EEG data will be align according to the onset of the cue and averaged across trials at each time point to obtain the movement related cortical potential curves. Peak amplitudes will be compared before and after the 10 sessions of active stimulation and before and after the 10 sessions of placebo stimulation using permutation based statistics.
Resting-state functional Magnetic Resonance Imaging (rs-fMRI) | Measured one time per day, at the days 2, 13, 14, and 25.
  In addition, the fMRI during rest will be used to analyze the connectivity between motor-related. Changes in connectivity will be explored and measured by calculation of global correlation, local correlation, amplitude low-frequency fluctuations, intrinsic connectivity and fractional amplitude low-frequency fluctuations. In addition, a seed-based analysis will be performed to check for changes in connectivity between the area of stimulation and other motor areas: M1, SMA, cerebellum and basal ganglia.
Voxel-based morphometry | Measured one time per day, at the days 2, 13, 14, and 25.
  Voxel-based morphometry is a proxy of gray matter concentration changes based on T1-weighted MRI. This will be evaluated in response to active and placebo stimulation. A flexible factorial design will address potential changes in grey matter after the stimulation. The investigators hypothesize that changes in gray matter will be observed for the stimulated region and functionally connected areas as M1, contralateral PMC, SMA, cerebellum and basal ganglia.
Brain-derived neurotrophic factor (BDNF) in serum | Measured twice per day, at the days 3, 12, 15 and 24. The first measure occurs before the intervention and the second measure after the intervention.
  Serum BDNF is proposed as a marker of plasticity mechanisms. Previous studies suggest that BDNF can be modulated by multiple-session rTMS protocols. However, no study has explored changes in BDNF after excitatory rTMS protocols in stroke participants. The investigators expect a higher change in BDNF levels after active stimulation in comparison with after placebo.

OTHER OUTCOMES:
Adherence | Through study completion, for 25 days.
  Number of missed sessions per participant
Upper extremity motor activity log (UE-MAL) | Measured one time per day, at days 2, 13, 14, and 25.
  The UE-MAL is a questionnaire that inspects how much and how well the participant uses their paretic arm during activities of daily living. Participants are asked standardized questions about how often they use their more-affected arm for different activities (Amount Scale or AS) and the perceived quality of their movements when executing such tasks (How Well Scale or HW). The evaluations are done on a scale from 0 to 5. 0 represents non-use and 5 is use equal to the non- paretic hand. The scores' explanations are printed on separate sheets of paper and are placed in front of the participant during the test administration. The sums of values recorded before and after the stimulation periods will be fed into an unpaired sample t-test to evaluate carryover effects whereas the differences observed between recordings before and after the stimulation will be fed into an unpaired sample t-test for the evaluation of initial evidence of the effect of rTMS.
Withdrawal rate | Through study completion, for 25 days.
  The proportion of participants that drop out.
Last item of the stroke impact scale (SIS) | Measured once per day, at days 2, 13, 14, and 25.
  The last item of the SIS will be used to ask participants to rank of their expected improvement due to the intervention from 0 to 100. This assessment will be used also after stimulation to assess the perceived improvement. The sums of values recorded before and after the stimulation periods will be fed into an unpaired sample t-test to evaluate carryover effects whereas the differences observed between recordings before and after the stimulation will be fed into an unpaired sample t-test for the evaluation of initial evidence of the effect of rTMS.
Micro fractional anisotropy (micro-FA) | Measured once per day, at days 2, 13, 14, and 25.
  Micro-FA is a proxy of white matter integrity that in contrast with FA can resolve ambiguities caused by crossing fibers. Micro-FA values will be obtained by acquiring diffusion-weighted images with a free waveform encoding pulse sequence. The micro-FA will be evaluated in the area of stimulation and areas that show changes in FA, in order to further characterize micro-structural arrangements elicited by the brain stimulation. A second-order cumulative model will be implemented for analysis.
Glial fibrillary acidic protein (GFAP) | Measured twice per day, at the days 3, 12, 15 and 24. The first measure occurs before the intervention and the second measure after the intervention.
  GFAP will be explored as it is proposed to change with plasticity due to the transient swelling of astrocytes during structural neuronal plasticity. The investigators expect a higher change in GFAP levels after active stimulation in comparison with after placebo.
Neurofilaments (light chain) | Measured twice per day, at the days 3, 12, 15 and 24. The first measure occurs before the intervention and the second measure after the intervention.
  Neurofilament light chains in blood will be inspected as they have been proposed as a marker of recovery after stroke. The investigators expect a higher change in Neurofilaments levels after active stimulation in comparison with after placebo.
Beta-synuclein | Measured twice per day, at the days 3, 12, 15 and 24. The first measure occurs before the intervention and the second measure after the intervention.
  Beta-synuclein will be explored because it has been proposed as a marker of synaptic alterations. The investigators expect a higher change in Beta-synuclein levels after active stimulation in comparison with after placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Flores-Sandoval, MsC, Study Chair — Charité Universitätmedizin Berlin and Max Planck Institute for Human Cognitive and Brain Sciences; Arno Villringer, MD PhD, Study Director — Max Planck Institute for Human Cognitive and Brain Sciences; Bernhard Sehm, PD. med., Principal Investigator — Max Planck Institute for Human Cognitive and Brain Sciences and Halle University; Vadim Nikulin, PhD., Principal Investigator — Max Planck Institute for Human Cognitive and Brain Sciences
Locations (1):
- Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will require approval by the local ethics committee (EC) of the researcher requesting the data along with public registration of the study. Data sharing will also be subject to compliance with the European Union General Data Protection Regulation.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After the end of the study and for 10 years
Access Criteria: The purpose for requesting the data and planned analysis must comply with the General Data Protection Regulation as well as Medical device regulation of the European Union.

REFERENCES:
- [Background] Tang Z, Han K, Wang R, Zhang Y, Zhang H. Excitatory Repetitive Transcranial Magnetic Stimulation Over the Ipsilesional Hemisphere for Upper Limb Motor Function After Stroke: A Systematic Review and Meta-Analysis. Front Neurol. 2022 Jun 20;13:918597. doi: 10.3389/fneur.2022.918597. eCollection 2022. PMID 35795793
- [Background] Peng Y, Wang J, Liu Z, Zhong L, Wen X, Wang P, Gong X, Liu H. The Application of Brain-Computer Interface in Upper Limb Dysfunction After Stroke: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Hum Neurosci. 2022 Mar 29;16:798883. doi: 10.3389/fnhum.2022.798883. eCollection 2022. PMID 35422693
- See also: Study webpage — https://www.cbs.mpg.de/study-applications/fgnme/innovative-neurotechnology-stroke